CLINICAL TRIAL: NCT02753166
Title: Dexamethasone as an Immediate Intervention to Reduce Long-Term Stress Responses
Brief Title: Dexamethasone as an Immediate Intervention
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15-01318
Record Dates: First submitted 2016-04-26; First posted 2016-04-27 (Estimated); Last update posted 2017-12-14 (Actual); Status verified 2017-12

CONDITIONS: Trauma
Keywords: PTSD (Post Traumatic Stress Disorder); Emergency Department
MeSH Terms: conditions — Wounds and Injuries; Combat Disorders; Emergencies | interventions — Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dexamethasone (Experimental)
  Interventions: Drug: Dexamethasone
- Control (No Intervention)

INTERVENTIONS:
Drug: Dexamethasone — After six (6) hours of the accident, subject will take 5 mg of DEX in the Emergency Department (ED). Within twenty-four (24) hours, the subjects will send in a saliva sample. After sexen (7) days, subjects will participate in a phone interview. After thirty (30) days, subjects will participate in an online assessment and return for a one month follow-up visit. Subjects will then participate in online assessments at months 3,6,9, and 12 months.
  Other Names: DEX
  Arms: Dexamethasone

SUMMARY:
To determine if a single dose of dexamethasone (5 mg) administered in the first 12 hours following a potentially traumatic event alters a) cortisol and FKBP5 RNA the next day in the periphery measured in saliva; b) FKBP5 methylation by 1 month; c) executive functioning and emotion regulation functioning; d) psychophysiological (heart rate, respiration, skin conductance) in response cued reminders of the trauma; e) enhances the likelihood of remission of PTSD symptom severity.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18-70 years
* Evidence of acute Post Traumatic Event (PTE) exposure defined by Diagnostic and Statistical Manual criterion 'A'
* Evidence of a significant stress response defined by DSM V PTSD criterion 'B' and meeting at least criteria for 'partial PTSD' or a minimum of 3 of 4 DSM V PTSD symptom criterion
* Score of 60 or higher on the Subjective Units of Distress Scale (SUDS)
* Living in New York tri-state area
* Fluency in English, Spanish

Exclusion Criteria:

* Admission to an intensive care unit or other overnight admission
* In the Emergency Department for more than 6 hours
* Evidence of ongoing traumatic exposure (e.g. domestic violence)
* Evidence of psychotic symptoms
* Evidence of homicidality/suicidality
* Adults with an open head injury, a positive CT scan, loss of consciousness >30 seconds or survivors in a coma
* Adults in police custody or Department of Correction (DOC) patients
* Inability to understand the study's procedures, risks, or side effects, or otherwise unable to give informed consent.
* Females who are nursing or pregnant (as confirmed by a positive urine pregnancy test).
* Permanent cardiac pacer implant.
* . Self-reported medical conditions that may be affected by DEX including asthma, epilepsy,diabetes, liver disease, kidney disease, thyroid disorder, muscle disorder, history of malaria,tuberculosis, osteoporosis, glaucoma or cataracts.
* Self-reported adverse reactions to steroids

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-12-12 (Actual); Study Completion 2017-12-12 (Actual)

PRIMARY OUTCOMES:
Change in score on PTSD symptom severity measured with the PTSD Check-List 5 (PCL-5) | 1 month, 3 months, 6 months, 9 months, and 12 months
  Mean symptom severity on the PCL-5 will be compared between groups using an independent samples T-test.

SECONDARY OUTCOMES:
Cortisol Levels measured from saliva samples | 24 hours post ED departure
Score on Subjective Units of Distress (SUDS) | 1 month, 3 months, 6 months, 9 months, and 12 months
  Scale of 0 to 10 for measuring the subjective intensity of disturbance or distress currently experienced by an individual. The individual self assesses where they are on the scale.
Score on the Kessler 6 Scale | 1 month, 3 months, 6 months, 9 months, and 12 months
  Measure of Psychological distress in the anxiety-depression spectrum
Score on Life Satisfaction Scale | 1 month, 3 months, 6 months, 9 months, and 12 months
  The Satisfaction with Life Scale to assess satisfaction with people's lives as a whole. The scale does not assess satisfaction with specific life domains, such as health or finances, but allows subjects to integrate and weigh these domains in whatever way they choose.
Score on Center for Epidemiologic Studies Depression Scale (CES-D) | 1 month, 3 months, 6 months, 9 months, and 12 months
Score on Perceived Ability to Cope with Trauma Scale (PACT) | 1 month, 3 months, 6 months, 9 months, and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Isaac Galatzer-Levy, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University Medical Center, New York, New York, United States